CLINICAL TRIAL: NCT03724279
Title: Safety and Effectiveness of ByCross Rotational and Aspiration Device for Revascularization of Total or Sub-total Occluded Peripheral Arterial Vessels of Luminal Diameter Equal to or Larger Than 3mm: A Prospective, Multi-center Study
Brief Title: Crossing Atheroma or Thrombus With ByCross Device for Revascularization of Peripheral Arteries of Diameter ≥ 3mm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taryag Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QA 213.06; U1111-1222-4481 (Registry Identifier: World Health Organization (WHO-UTN)); DRKS00015758 (Registry Identifier: German Clinical Trials Registrar (DRKS))
Record Dates: First submitted 2018-10-17; First posted 2018-10-30 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Arterial Occlusive Diseases
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Thrombectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ByCross Atherectomy and Thrombectomy (Experimental): Percutaneous intervention including ByCross atherectomy and Thrombectomy potentially followed with PTA and/or stent placement
  Interventions: Device: ByCross Atherectomy and Thrombectomy

INTERVENTIONS:
Device: ByCross Atherectomy and Thrombectomy — After assessment of the lesion by angiography the ByCross is advanced over a 0.035" guidewire through a sheath to the occlusion. Activation will rotate the shaft and start aspiration. Under fluoroscopy the ByCross is advanced continuously over the wire. in case passage is not possible the ByCross tip is advanced into the occlusion for 10mm, then wire is advanced to check is passage is possible, this is repeated until passage by the wire is achieved. At harder lesion the speed is set to high. Once the occlusion is crossed the ByCross tip is enlarged, device is advanced once more to increase opening. Additional adjunctive treatment may be performed per physician's discretion and according to standard of care. Performance criteria of the intervention is to achieved more than 70% opening.

SUMMARY:
The aim of the study is to demonstrate safety and effectiveness of ByCross Rotational and Aspiration device used for revascularization of total or sub-total occluded peripheral arterial vessels equal to or larger than 3mm in diameter.

The ByCross is a single use, disposable, minimal invasive aspiration rotational atherectomy device. The ByCross is aimed to enable effective revascularization and restore blood flow in peripheral occluded vessels. In cases that the artery is completely blocked such that opening is not possible with currently available solutions and the procedure cannot be completed, the device is capable of crossing the blocked lesion without guiding wire and enables the completion of the procedure in a safe and effective manner, thus potentially eliminating the need for open bypass surgery. The ByCross can be used in several pathologies: calcified atheroma, old and fresh thrombus.

Eligible adult patients with symptoms due to chronic sub-total and total occlusion will be enrolled and undergo percutaneous procedure including use of ByCross which will normally be followed by balloon inflation (Percutaneous Transluminal Angioplasty) in the artery at location where blockage has been opened by ByCross to further open the artery and restore full opening, and in some case followed by placement of a stent for long term stabilization.

For demonstrating safety and effectiveness up to 42 patients will be enrolled. the procedure will take up to 2 hours followed by up to 48 hour hospitalization. Patients will then come for follow-up monitoring and examination 30 days and 6 months after procedure. Although this is unlikely, in some cases the physician can decide during procedure that following ByCross opening of the artery, ballooning or stent is not required. In this case the patient will come for another follow-up visit after 12 month.

DETAILED DESCRIPTION:
Occlusive vascular disease (OVD) is the leading cause of mortality and morbidity in the Western world. Arterial obstructions generally start as a build-up of harder atherosclerotic material on which clotted blood (thrombus) forms, whereas veins obstruction contains mostly thrombus. Over 10 million patients in the US suffer from peripheral arterial disease (PAD) including 750,000 critical limb ischemia patients who are at risk of limb amputation.

The existing pharmacological and bypass surgical methods to treat OVD are risky, expensive, and time-consuming. Overcoming these shortcomings presents a substantial opportunity for a mechanical catheter. Atherectomy with mechanical catheters has been used clinically for many years, and by now the clinical outcome of atherectomy is known as reflected by multiple clinical studies. The potential benefit of the technique compared with percutaneous transluminal angioplasty (PTA) and/or Stenting alone or as an adjunctive therapy has also been discussed, and more recently as an adjunctive prior to PTA with a drugeluting balloon and stenting. The existing catheters designed mainly for arteries are expensive, complicated to operate, demonstrate limited reduction in level of stenosis, might cause perforations, distal embolization and hemolysis, have no or poor aspiration, and cannot cross occlusions without passage of guidewire first. Despite the common use of these therapies and current benefits, there remain significant opportunities to extend catheter-based treatments with improved outcomes, to more patients and at lower cost.

The ByCross is a minimal invasive, single use atherectomy and thrombectomy device, which is introduced over the wire into the peripheral vasculature for revascularization of chronic occluded peripheral vessels. The ByCross has a coaxial flexible rotating shaft with an expandable tip and integrates an independent aspiration system for suction of thrombotic material. The expandable tip is an elastic arc that can bow and enlarge the tip diameter from external tip diameter of 1.7mm at closed condition to 4.7mm at open condition. As the shaft rotates, the tip breaks the calcified atheroma or thrombus into small particles, which are simultaneously aspired into the shaft and removed into the attached collection bag. The ByCross allows injection of contrast medium and thrombolytic agents through the rotating tip during the procedure for continuance imaging and prevention of appositional thrombus formation. Due to its no-symmetrical helical design the tip rotation is eccentric, causing the tip to recenter is self within the lumen as it rotates. While ByCross is introduced over a guide wire, it does not require the passage of an occlusion with the wire first. To cross the occlusion the ByCross is advanced with running motor forth and back in a closed condition. Once the occluded segment is crossed the procedure is repeated with open tip at larger diameter vessels to further remove the remaining atheroma or thrombus. The ByCross is battery powered, and includes a remote-control unit which allows the user full ergonomic control of the device next to the puncture site.

Based on compliance with standard requirements, design process and risk analysis process. The risk of occurrence of adverse events is not expected to be greater than the risk reported for other devices available in the market today. More over the past animal test supports the expected low risk. This study, aside to performance investigation, is intended to validate this. The potential significant advantage of the ByCross device in the treatment of chronic limb ischemia is the ability to cross Chronic Total Occlusion (calcified atheroma and/or thrombus, in oppose to other atherectomy devices which can only cross partial occluded vessel due to the necessity of progressing over the wire). Thus, instead of aborting the procedure, completion of revascularization procedure percutaneously is possible. In addition, the ByCross enables, due to its design, to achieve superior patency, injection of contrast medium and antiplatelet during operation of the radio-opaque tip, and enables simultaneous aspiration.

These benefits potentially reduce prolonged percutaneous procedures if other means are required to enable chroni total occlusion (CTO) passage by guidewire, and, might, in the future, reduce the number of bypass surgeries in peripheral arteries, all with no risk compared to long term clinical use of equivalent devices.

Information gathered in this study will further assure the ByCross device as superior solution enabling more beneficial minimal invasive procedure for the subjects with the same indication for treatment.

The study is multi-center, single arm, open label, prospective study. 42 patients with total or subtotal occlusion at target vessel bearing length equal to or larger than 3cm at vessels diameter of 3mm or larger will be enrolled to the study. Eligible consented subjects will undergo a procedure and treated with the ByCross device. Additional adjunctive treatment (such as PTA, stenting etc.) may be performed per physician's discretion and according to standard of care. Assessment of device safety and performance will be performed intra and post procedural, at discharge, at 30 days post procedure and at 6 months. Subjects that will undergo procedure using ByCross only with NO adjunctive therapy will be followed-up at 12 months as well. The overall duration of participation for each subject is expected to be up to 7 months and 13 months for those that undergo procedure using ByCross only.

Primary outcome measures are divided into two: performance and safety. The null hypotheses will be tested via the lower limit of the one-sided 95% exact confidence interval for the respective proportions. The expected Acute Procedural Success rate is 95% as is the rate of subjects free of device-related Major Adverse Events (MAEs) throughout a 30-day follow-up. The sample size required to achieve a lower one-sided 95% exact confidence limit that is greater than 85%, if the point estimate of the proportion is 95%, is calculated as 40 patients. To accommodate a potential 5% drop-out prior to completing 30 days follow-up, up to 42 patients may be required to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Subject has documented symptomatic (Rutherford 2-6), chronic peripheral vascular disease requiring percutaneous intervention and are indicated for atherectomy at superficial femoral (SFA) and/or popliteal artery and/or tibioperoneal trunk (TPT).
* Target lesion is at least 10mm distal to the SFA origin and at least 10mm proximal to the distal end of the TPT.
* Total or sub-total occlusion of target vessel (stenosis ≥80%)
* Vessel lumen ≥3.0mm
* Lesion length ≥3.0cm
* Subject has been informed on the nature of the study and is willing and able to provide informed consent
* Subject is capable of meeting study requirements including presences at follow-up visits

Exclusion Criteria:

* Subject is unable to take antiplatelet drugs
* Vessel of the cardiopulmonary, coronary or cerebral circulation
* Subject has anticipated life expectance < 12 month
* Subject is diagnosed with impaired renal function (creatinine >2.5 mg/dL)
* Subject has undergone or planned surgical or endovascular procedure 15 days before or after the study procedure
* Vessel lumen <3.0mm
* Stent at access and target vessel or In-stent restenosis at target lesion
* Target and/or access vessel include by-pass graft
* Target vessel is dissected
* Target is at vessel segment which includes tortuous course with radius of curvature <= 40mm
* Access pathway includes tortuous course with radius of curvature <= 25mm
* Target and/or access vessel includes aneurysm altered segments
* Persistent vasospasm
* Known or suspected allergy to any of the components of the sys-tem or to a medicinal product to be administered in connection with the planned procedure
* Subject is pregnant or planning to become pregnant within the study period, or lactating mothers
* Subject is enrolled to another clinical investigation that might interfere with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Rate of subjects with post atherectomy stenosis ≤ 50% and post procedure stenosis ≤ 30% | Up to 8 hours post-procedure
  Passage of the occlusion by the ByCross device and post atherectomy residual stenosis (assessed using angiograph) ≤ 50% to allow for angioplasty and/or stenting if required, and complete procedural success of residual stenosis ≤ 30%, with no Serious Adverse Events (SAE) during the procedure
Rate of major adverse events | 30-days follow-up
  Major Adverse Events (MAE), at 30 days follow-up. Each Major Adverse Event (MAE) will be assessed to determine whether its root cause is device-related complication, adjunctive therapy (e.g balloon and/or stent) related complication or other related complication.

SECONDARY OUTCOMES:
Stenosis level | up to 96 hours, 30-days and 6-months follow-up
  No deterioration in target vessel stenosis level at 30 and 6 months compared to post procedure level. Stenosis evaluated using Duplex Ultrasound.
Ankle Brachial Pressure Index | up to 96 hours, 30-days and 6 months follow-up
  Ankle Brachial Pressure Index (ABPI) at hospital discharge, 30 days and 6 months follow-up.
  ABPI is the ratio between the systolic blood pressure of the ankle divided by the systolic blood pressure of the arm. Scale can be larger than 0 and smaller than 1.2. 0.9-1.4 range indicates normal condition while values smaller than 0.8 indicates peripheral vascular disease. Lower value indicates higher severity. Scale higher than 1.4 indicates distortion of measurements due to abnormal vessel behavior (e.g. hardening).
Major adverse events | Up to 8 hours post-procedure, up to 96 hours, 6-months follow-up, and 12-months if applicable
  Major Adverse Events (MAE) during procedure, at hospital discharge at 6 months follow-up for all patients, and at 12 months follow-up for subjects that undergo procedure using ByCross with NO adjunctive therapy. Each Major Adverse Event (MAE) will be assessed to determine whether its root cause is device-related complication, adjunctive therapy (e.g balloon and/or stent) related complication or other related complication.

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Tessarek, M.D., Principal Investigator — Bonifatius Hospital Lingen
Locations (2):
- Germany (2):
  - Augusta-Krankenhaus, Düsseldorf
  - Bonifatius Hospital Lingen, Lingen

REFERENCES:
- [Derived] Tessarek J, Kolvenbach R. Safety and effectiveness of bycross rotational atherectomy and aspiration device: a prospective, multi-center pre-market approval study. CVIR Endovasc. 2023 Mar 29;6(1):19. doi: 10.1186/s42155-023-00363-0. PMID 36988757